CLINICAL TRIAL: NCT06559514
Title: The Effectiveness of Group-based Multi-Component Psycho-Educational Interventions (GMC-PEIs) on Burden, Depression, Coping and Quality of Life in Communication Partners of Older Adults With Hearing Impairment
Brief Title: Effect of Psycho-Educational Interventions in Communication Partners of Older Adults With Hearing Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202304022RINA
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Older Adults; Hearing Impairment; Nursing; Communication Partners
Keywords: group-based multi-component interventions; psychoeducation; hearing impairment; older adults; communication partners; burden; depression; coping; quality of life
MeSH Terms: conditions — Hearing Loss; Depression

STUDY DESIGN:
Intervention Model Description: In this single-blind, randomized controlled trial, adults aged years or older living with hearing impairment elderly will be randomized into either the intervention group (group-based multi-component psychoeducational inventions, GMC-PEIs intervention group) or the control group (waitlist control group).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-based multi-component psycho-educational inventions (GMC-PEIs) (Experimental): Group-based multi-component psycho-educational interventions. The participants were randomly assigned to either the experimental group or the waiting-list control group, using a computer-generated list of random numbers.
  Interventions: Behavioral: Group-based multi-component psychoeducational inventions (GMC-PEIs)
- Controls group (No Intervention): Waitlist control group

INTERVENTIONS:
Behavioral: Group-based multi-component psychoeducational inventions (GMC-PEIs) — The participants were randomly assigned to either the experimental group, using a computer-generated list of random numbers.
  Arms: Group-based multi-component psycho-educational inventions (GMC-PEIs)

SUMMARY:
Hearing impairment is a critical health problem throughout the world. In addition, having an impact on the biopsychosocial functioning of older adults, it places enormous stress and burden on communication partners who interact with older adults with hearing impairment every day. These communication partners generally have restrictions to their social lives and an increased communication burden, as well as symptoms of depression and adopting maladaptive coping and poorer quality of life. Therefore, group-based multi-component psycho-educational interventions are recommended. The purposes of this study are to examine the effects of group-based multi-component psycho-educational interventions (GMC-PEIs) on burden, depression, coping and quality of life in communication partners of older adults with hearing impairment. The single-blind, randomized control trial will include communication partners of older adults with hearing impairment. Participants will be randomized to either intervention groups or control groups.

DETAILED DESCRIPTION:
The study will be an experimental design featuring repeated measures, with data collected from a pretest, a posttest and a follow-up test. An estimated total of 92 participants will be randomly assigned to experimental and control groups. The experimental group will participate in a 6-week group-based multi-component psycho-educational interventions (GMC-PEIs), including provide information on communication skills training, clear speech training, psychosocial support, stress management and successful person testimonial, consisting of 60-minute sessions once per week, while the control group will be put on a waiting-list group. Each group will be assessed of the outcomes at 3 time points: baseline (T0), three months following the intervention (T1) and again at six months following the intervention (T2). The investigators will use the Significant Other Scale for Hearing Disability (SOS-HEAR), the 10-item version of the Center for Epidemiological Studies Depression Scale (10-Item CES-D), the Brief Coping Orientation to Problems Experienced Scale (B-COPE), the Short Form Health Survey (SF-12) and the International Outcome Inventory for Hearing Aids-Significant Other (IOI-HA-SO) as the outcome indicators. The principle of intention-to-treat (ITT) analysis will be used, and the result will be analyzed mainly by generalized estimating equation (GEE).

ELIGIBILITY:
Inclusion Criteria:

* being18 or older
* living with older adults with hearing impairment
* they were indicated that as primary communication partner
* no known hearing loss
* having normal cognitive function
* articulate in the Mandarin Chinese language
* signing a consent form to participate

Exclusion Criteria:

* severe psychiatric disorders
* the communication partner who is hired as a caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline the Significant Other Scale for Hearing Disability, at 3 months, and 6 months. | baseline, 3th, 6th month
  A score of participants in baseline burden as assessed by the Significant Other Scale for Hearing Disability. The overall score ranging from 0 to 108, which higher scores indicating higher severe burden.
Change from baseline the 10-item version of the Center for Epidemiological Studies Depression Scale at 3 months, and 6 months. | baseline, 3th, 6th month
  A score of participants in baseline depression as assessed by the 10-item version of the Center for Epidemiological Studies Depression Scale. The overall score ranging from 0 to 30, which higher scores indicating severe depression.
Change from baseline the Brief Coping Orientation to Problems Experienced Scale at 3 months, and 6 months. | baseline, 3th, 6th month
  A score of participants in baseline coping as assessed by the Brief Coping Orientation to Problems Experienced Scale. The overall score ranging from 0 to 100, which higher scores indicating better coping.
Change from baseline the Short Form Health Survey(SF-12) at 3 months, and 6 months. | baseline, 3th, 6th month
  A score of participants in baseline quality of life as assessed by the Short Form Health Survey(SF-12) . The overall score ranging from 0 to 100, which higher scores indicating better quality of life.
Change from baseline the International Outcome Inventory for Hearing Aids-Significant Other at 3 months, and 6 months. | baseline, 3th, 6th month
  A score of participants in baseline overall intervention effectiveness and hearing aids satisfaction as assessed by the International Outcome Inventory for Hearing Aids-Significant Other. The overall score ranging from 7 to 35, which higher scores indicating better effectiveness of the intervention and aids satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Meei-Fang Lou, Principal Investigator — School of Nursing, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, No. 1, Sec. 1, Jen-Ai Rd., Taiwan

IPD SHARING:
Plan to Share IPD: No